CLINICAL TRIAL: NCT04289441
Title: "Randomized Controlled Double-blind Trial With Lactobacillus Salivarius LS01 (DSM 22775) and Bifidobacterium Breve B632 (DSM 24706) for Paediatric Asthma Management"
Brief Title: Probiotics in Paediatric Asthma Management
Acronym: ProPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probiotical S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCCE n.41486
Record Dates: First submitted 2020-01-23; First posted 2020-02-28 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: Randomized controlled double-blind trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic treatment (Active Comparator): For the first 8 weeks was administered 1 sachet in the morning and 1 in the evening, for the last 8 weeks was administered 1 sachet per day
  Lactobacillus salivarius LS01 (DSM 22775): 10^9 CFU Bifidobacterium breve B632 (DSM 24706): 10^9 CFU Maltodextrin and silicon dioxide
  Interventions: Dietary Supplement: Bifiasthm
- Placebo treatment (Placebo Comparator): For the first 8 weeks was administered 1 sachet in the morning and 1 in the evening, for the last 8 weeks was administered 1 sachet per day
  Maltodextrin and silicon dioxide
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifiasthm — Subjects will be instructed to take an active or placebo sachet twice daily for eight weeks, and subsequent intake of one dose daily for a further eight weeks.
  Arms: probiotic treatment
Dietary Supplement: Placebo — Placebo
  Arms: Placebo treatment

SUMMARY:
Randomized controlled double-blind trial in a child population with allergic asthma and recurring wheezing, undergoing probiotic treatment with Bifiasthm with the aim of assessing the reduction in asthma attacks.

DETAILED DESCRIPTION:
Allergic disorders have dramatically increased in prevalence over the past decade, particularly in developed countries, and primary prevention of allergic disease has proved an elusive goal. There is increasing evidence that the airway microbiome influences the development of wheezing and childhood asthma. Probiotics are increasingly considered as a promising treatment for the correction of dysbiosis, reduction of systemic inflammation, and modulation of allergic diseases. The aim of this study is, therefore, to evaluate the efficacy of Bifidobacterium breve B632 (DSM 24706) and Lactobacillus salivarius LS01 (DSM 22775) in the prevention of asthmatic allergies in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* The study will include all children aged 6 to 14, with slight and moderate persistent asthma according to GINA 2015 criteria (asthma classification did not change in GINA 2015 and 2016 guidelines), whether or not showing positive skin allergometric tests, as well as all children aged 2 yrs, 364 days to 5 years, 364 days, with recurring wheezing, whether or not diagnosed with asthma (positive and/or negative prick).

Exclusion Criteria:

* Severe persistent asthma
* Known congenital or acquired immunodeficiencies
* Cystic fibrosis
* Chronic pulmonary diseases (bronchodysplasia)
* Age < 1 yr, 364d and 14 yrs

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Reduction in Asthma episodes | 12 months
  Reduction in the frequency and severity of asthma crises, the evaluation is performed using Guidelines for management of Asthma, Italian Society of Pediatricians
Reduction in wheezing | 12 months
  Reduction in the frequency of wheezing episodes, numerical evaluation.

SECONDARY OUTCOMES:
Reduction of adminstrated drug quantity | 12 months
  Reduction in the administered drug quantity for asthma crisis treatment
Reduction in treatment time | 12 months
  use of short-term treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Ambulatory, Pozzuoli, Naples, Italy

REFERENCES:
- [Derived] Ciprandi G, Schiavetti I, Cioffi L, Pane M, Drago L. The Probiotics in Pediatric Asthma Management (PROPAM) study: A Post Hoc analysis in allergic children. Ann Allergy Asthma Immunol. 2022 Jul;129(1):111-113. doi: 10.1016/j.anai.2022.04.026. Epub 2022 Apr 26. No abstract available. PMID 35487387